CLINICAL TRIAL: NCT06420024
Title: Acceptance and Commitment Therapy (ACT) for Older Adults Who Hear Voices: a Hermeneutic Single-case Efficacy Design (HSCED) Series
Brief Title: ACT for Older Adults Who Hear Voices (HSCED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government); Derbyshire Healthcare NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23007
Record Dates: First submitted 2023-03-23; First posted 2024-05-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-08

CONDITIONS: Hearing Voices When No One is Talking
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Hermeneutic Single Case Efficacy Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participant will receive ACT intervention
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — See: https://link.springer.com/chapter/10.1007/0-306-48581-8_1

SUMMARY:
Hearing voices (often referred to as "auditory hallucinations") is a common experience amongst the older adult population (those 65+ years of age) and can be associated with increased psychological distress. Acceptance and Commitment Therapy (ACT) is a psychological therapy that aims to reduce distress of hearing voices by altering the relationship someone has with voices, and has been shown to improve distress levels for working age adults who hear voices. ACT also appears to be a suitable intervention for older adults distressed by hearing voices, however, there is currently no research that has examined this. Therefore, research is now needed to evaluate whether ACT can support older adults who experience distress from hearing voices.

This study will use a case study based research method, known as a Hermeneutic Single-Case Efficacy Design (HSCED) series. This method will involve 3 participants who will receive ACT for hearing voices. This will be delivered across approximately twelve 90-minute sessions. Participants will be asked to complete measures that assess areas such as distress levels and quality of life, which will be completed before, during and after therapy. A detailed report of each participant's level of progress will then be generated and evaluated by expert judges. This will determine whether progress has occurred as a direct result of the therapy, or due to other reasons, and allow conclusions to be drawn about the use of ACT for older adults distressed by hearing voices.

Participants will be recruited from either Local Mental Health Teams at Nottinghamshire NHS Foundation Trust, or from the Hearing Voices Group in Beeston (Nottingham). Participants will be required to be age 65+ years and currently experience hearing voices that cause them distress.

This study will be funded by the NHS and is estimated to last approximately 12-months with 5-months of participant involvement.

DETAILED DESCRIPTION:
Chief Investigator:

Dr Danielle De Boos

Objectives:

To investigate the efficacy of Acceptance and Commitment Therapy for older adults who hear voices in a Hermeneutic Single-Case Efficacy Design series.

Trial Configuration:

Case study series, recruited from multiple centres.

Settings:

Secondary care older adult mental health service and charity-based support groups.

Sample size estimate:

3

Number of participants:

Three participants. If a participant withdraws, a replacement participant will be sought.

Eligibility criteria:

Individuals who are 65+ years of age, experience moderate levels of distress (as defined by the Depression, Anxiety and Stress Scales-21), have capacity to provide informed consent, and express willingness to engage in the intervention are eligible to participate providing they do not have a diagnosis of dementia/cognitive impairment, are not currently receiving other psychological therapy and are able to independently communicate in English.

Description of interventions:

Acceptance and commitment therapy adapted to suit the needs of older adults. Twelve sessions are expected to take place, with a review at session six.

Duration of study:

Up to 20 months.

Outcome measures:

Personal Questionnaire (simplified) will be reviewed weekly.

At baseline, pre-therapy, mid-therapy, post-therapy, and follow-up (4-6 weeks) participants will complete the following outcome measures:

* Voices Acceptance and Action Scale-9,
* Beliefs about voices questionnaire-revised,
* Depression, Anxiety and Stress Scales-21,
* Comprehensive assessment of Acceptance and Commitment Therapy processes (short-form),
* Older People's Quality of Life questionnaire (brief version),
* Psychotic Symptom Rating Scale (Auditory Hallucination sub-scale).

Participants will also complete a change interview post-therapy with Trainee Clinical Psychologist (Jennifer Welch; University of Nottingham / University of Lincoln) who is independent to this study.

Statistical methods:

Reliable Change Index; adjudication panel; Framework Analysis; correlations; visual analysis

ELIGIBILITY:
Inclusion Criteria:

* Currently experiences HV
* 65+ years of age
* Moderate levels of distress. This will be measured using recommended "Moderate" severity level cut-off scores on the Depression, Anxiety and Stress Scales-21 (Lovibond & Lovibond, 1995) following the completion of Informed Consent Forms.
* Having capacity to provide informed consent (in accordance with the Mental Capacity Act)
* Willingness to engage in the intervention

Exclusion Criteria:

* Diagnosis of cognitive impairment or dementia (based on self-report), as this indicates a degree of cognitive impairment that would be difficult to accommodate for.
* Current engagement with another psychological therapy
* Unable to independently communicate in English without an interpreter (based on researcher's discretion at recruitment).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Voices Acceptance and Action Scale-9 (Brockman et al., 2015) | Approx. 0 weeks (baseline), 6 weeks (mid-therapy), 12-14 weeks (post therapy), 16-18 weeks (4-6 week follow-up) following enrolment to the study.
  Acceptance-based attitudes and actions in relation to voices
Beliefs about voices questionnaire-revised (Chadwick et al., 2000) | Approx. 0 weeks (baseline), 6 weeks (mid-therapy), 12-14 weeks (post therapy), 16-18 weeks (4-6 week follow-up) following enrolment to the study.
  Beliefs, emotions, and behaviours relating to auditory hallucinations.
Depression, Anxiety and Stress Scales-21 (Lovibond & Lovibond, 1995) | Approx. 0 weeks (baseline), 6 weeks (mid-therapy), 12-14 weeks (post therapy), 16-18 weeks (4-6 week follow-up) following enrolment to the study.
  Depression, Anxiety and Stress
Comprehensive assessment of Acceptance and Commitment Therapy processes, short-form (Morris et al., 2019) | Approx. 0 weeks (baseline), 6 weeks (mid-therapy), 12-14 weeks (post therapy), 16-18 weeks (4-6 week follow-up) following enrolment to the study.
  Psychological flexibility
Older People's Quality of Life questionnaire, brief version (Bowling et al., 2013) | Approx. 0 weeks (baseline), 6 weeks (mid-therapy), 12-14 weeks (post therapy), 16-18 weeks (4-6 week follow-up) following enrolment to the study.
  Quality of Life
The Psychotic Symptom Rating Scales (Haddock et al., 1999) - Auditory Hallucination Sub-Scale | Approx. 0 weeks, 6 weeks, 12-14 weeks, 16-18 weeks following enrolment to the study.
  Symptom severity of auditory hallucinations

SECONDARY OUTCOMES:
Simplified Personal Questionnaire (Elliott et al., 1999) | Weekly during the intervention (i.e., once per week during the intervention phase - this is anticipated to occur within the first 12-14 weeks of the participant's involvement with the study)
  Individualised client-generated goals

CONTACTS AND LOCATIONS:
Overall Officials: Danielle De Boos, DClinPsy, Study Chair — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Derbyshire Healthcare NHS Foundation Trust, Derby, Derbyshire
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No